CLINICAL TRIAL: NCT06195267
Title: Protective Effect of Sivelestat Against Negative Pulmonary Function and Organ Dysfunction After Cardiovascular Surgery (PANDA VI)
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANDA VI
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Aortic Dissection; Systemic Inflammatory Response Syndrome; Cardiovascular Diseases (CVD)
Keywords: Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Aortic Dissection; Systemic Inflammatory Response Syndrome; Cardiovascular Diseases | interventions — sivelestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sivelestat (Experimental)
  Interventions: Drug: Sivelestat
- Blank control (Sham Comparator): The control group did not receive any intervention.
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Sivelestat — The total 24-hour dose of Sivelestat sodium (4.8mg/kg) was dissolved with 50 ml normal saline. The drug flow rate was set at 2ml/h with an intravenous microinfusion pump, and the constant speed infusion was completed in 24h.
  Arms: Sivelestat
Drug: Blank control — Patients only received standard treatment and care.
  Arms: Blank control

SUMMARY:
Systemic inflammatory response syndrome (SIRS) and multiple organ dysfunction syndrome (MODS) are the major causes of death in patients with cardiovascular diseases. Therefore, the prevention of SIRS and MODS is of great clinical value, and immunomodulatory therapy with sivelestat may be beneficial. This study was designed to test the hypothesis that the administration of sivelestat during the acute phase of cardiovascular diseases will result in a reduced incidence of SIRS and MODS.

ELIGIBILITY:
Inclusion Criteria:

* The patients are conformed to 2010 ACC/AHA guidelines for the diagnosis and treatment of thoracic aortic disease (TAD) within two weeks of onset;
* Patients with type A acute aortic syndrome confirmed clinically and radiologically and planning to undergo emergency surgery were enrolled.
* The patients' age between 18 ~90 years old.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients allergic to sivelestat sodium;
* Lactating women and pregnant women;
* Patients with mental diseases, drug and alcohol dependence;
* Refuse to participate in this study and refuse to sign the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The highest SOFA score of 7 days after surgery | 7 days after surgery
  The daily SOFA score after baseline was calculated for each patient on the basis of five organ systems: cardiovascular, respiratory, renal, hepatic, and coagulation systems. (Scores for each system range from 0 to 4, with higher scores indicating more severe organ-system dysfunction).

SECONDARY OUTCOMES:
all-cause mortality | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Beijing
  - The First Affiliated Hospital of Nanjing Medical University and Jiang ye-fan, Nanjing

IPD SHARING:
Plan to Share IPD: Undecided